CLINICAL TRIAL: NCT01254461
Title: A Phase I, Open Label, Randomised, Parallel Group Study of Repeated Oral Doses of AZD1981 (100 mg Twice Daily and 400 mg Twice Daily Via Tablet) for Eight Days and Single Doses of Pravastatin (Pravachol® Tablet 40 mg) to Evaluate the Pharmacokinetic Interaction of AZD1981 and Pravastatin in Healthy Male Volunteers
Brief Title: A Drug-Drug Interaction Study Between AZD1981 and Pravastatin to Study the Effect of AZD1981 on the Kinetics of Pravastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Christer Hultquist/Medical Science Director, AstraZeneca R&D
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D9830C00016; 2010-023876-14 (EudraCT Number)
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Drug Interaction
Keywords: Phase 1; Drug-Drug interaction; pravastatin; AZD1981; The pharmacokinetics resulting from AZD1981 and pravastatin interaction; The effects of taking a combination of AZD1981 and pravastatin
MeSH Terms: interventions — AZD1981; Pravastatin

ARMS (2):
- A (Experimental)
  Interventions: Drug: AZD1981; Drug: pravastatin
- B (Experimental)
  Interventions: Drug: AZD1981; Drug: pravastatin

INTERVENTIONS:
Drug: AZD1981 — 100 mg per oral, twice daily for 8 days
  Arms: A
Drug: AZD1981 — 4x100 mg per oral, twice daily for 8 days
  Arms: B
Drug: pravastatin — 40 mg, once daily at Day 1, period A and Day 8, period B
  Other Names: pravachol

SUMMARY:
The primary purpose of this study is to determine whether the treatment with AZD1981 will affect the pharmacokinetics of pravastatin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18 to 55, inclusive
* Have a body mass index between 19 and 30 kg/m2 and weight at least 50 kg and no more than 100 kg, inclusive
* Be a non-smoker or ex-smoker who has stopped smoking for >6 months prior to screening
* Volunteers must be willing to use barrier methods of contraception during study and 3 months after the end of their participation in the study

Exclusion Criteria:

* Any clinically significant disease or disorder
* Any clinically relevant abnormal findings in physical examination

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics for pravastatin measured by Cmax and AUC | Pharmacokinetic (PK) sampling will be performed on Day 1, period A and on Day 7-8, period B
  Pharmacokinetics for pravastatin measured by Cmax and AUC

SECONDARY OUTCOMES:
AUC | PK sampling will be performed on Day 1, period A and on Day 7-8, period B
  Pharmacokinetics for pravastatin measured by AUC[0-t],Cmax (tmax), CL/F, t1/2λz, Vz/F, MRT
AUCτ | PK sampling will be performed on Day 7 and Day 8, period B
  Pharmacokinetics for AZD1981 measured by AUCτ,Css,max, Css, max (tmax ss), CLss/F, t1/2λz, Vz/F, MRT
Safety and tolerability | Safety will be monitored continously and safety assessments will be made on several occasions throughout the whole study
  Safety and tolerability of AZD1981

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Uppsala, Sweden